CLINICAL TRIAL: NCT02205151
Title: An Open-label, Randomized, Single-dose, 2×2 Crossover Study to Compare the Pharmacokinetics of Fimasartan/Amlodipine Combination Tablet and Coadministration of Fimasartan and Amlodipine as Individual Tablets in Healthy Male Volunteers
Brief Title: To Compare the Pharmacokinetics of Fimasartan/Amlodipine Combination Tablet and Coadministration of Fimasartan and Amlodipine as Individual Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Kyunghee university hospital A Drug Analytical Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BR-FAC-CT-101
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
Keywords: Fimasartan
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment AB (Other): Treatment A (1 day) → wash-out(14days) → Treatment B (1 day)
  Treatment A : Fimasartanm and Amlodipine
  Treatment B : Fimasartan/Amlodipine combination
  Interventions: Drug: Fimasartan; Drug: Amlodipine; Drug: Fimasartan/Amlodipine combination
- Treatment BA (Other): Treatment B (1 day) → wash-out(14days) → Treatment A (1 day)
  Treatment A : Fimasartanm and Amlodipine
  Treatment B : Fimasartan/Amlodipine combination
  Interventions: Drug: Fimasartan; Drug: Amlodipine; Drug: Fimasartan/Amlodipine combination

INTERVENTIONS:
Drug: Fimasartan
Drug: Amlodipine
Drug: Fimasartan/Amlodipine combination

SUMMARY:
An Open-label, Randomized, Single-dose, 2×2 Crossover Study to Compare the Pharmacokinetics of Fimasartan/Amlodipine Combination Tablet and Coadministration of Fimasartan and Amlodipine as Individual Tablets in Healthy Male Volunteers

DETAILED DESCRIPTION:
After subjects have signed informed consent voluntarily, they go through screening period for within 21 days.

As period I, subjects of A Group take fimasartan and amlodipine at 1st day and subjects of B Group take fimasartan/amlodipine combination at 1st day.

And then, after wash out for 14 days, as period II, subjects of A Group take fimasartan/amlodipine combination at 15th day and subjects of B Group take fimasartan and amlodipine at 15th day.

At each period, subjects of A Group have blood sampling 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 144 hour after medication(18 times in each period, 36 times in total).

At each period, subjects of B Group have blood sampling 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 144 hour after medication(18 times in each period, 36 times in total).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject, aged 19- 50 years at screening.
2. Body weight of ≥ 50 kg and within ± 20% of ideal body weight (IBW)(kg) = {height (cm) - 100} * 0.9
3. Subjects must be able to listen to and understand the detailed statement of informed consent, and willing to decide to participate in the study, follow the study directions and provide written informed consent

Exclusion Criteria:

1. History of gastrointestinal disease (i.g., Crohn's disease, active peptic ulcer) or resection operation that may affect the absorption of the study drug (excluding simple appendectomy or herniorrhaphy)
2. History of clinically significant hypersensitivity to study drug, any other drug or additives (yellow no.4).
3. Subject that is judged inappropriate for participating in the study based on physical examination
4. The levels of ALT(Aspartate Transaminase), AST (Alanin Transaminase) or total bilirubin > 1.5 x the upper limit of normal or eGFR < 60 mL/min/1.73m (calculated by MDRD)
5. Evidence of hereditary disease, including galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
6. systolic ≥ 140 mmHg or ≤ 100 mmHg, diastolic ≥ 90 mmHg or ≤ 65 mmHg), measured after taking a rest for 5minutes
7. Take any other study's investigational products within 90 days prior to the first administration of study drug
8. Donation of whole blood within 60 days prior to the first administration of study drug, or donation of any blood products within 30 days prior to the first administration of study drug
9. Intake food like Grapefruit juice (*e.g., Grapefruit juice ≥ 1L /day) within 7 days prior to administration of study drug
10. Use of any prescribed drugs or herbal remedies within 14 days, or use of any over-the-counter medication or vitamins within 7 days prior to the first administration of study drug
11. Positive serologic tests (HBsAg, HCV Ab, HIV Ag/Ab, VDRL)
12. Subject that is judged inappropriate for participating in the study by an investigator, based any other reason

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
(Cmax) | 0~144 hour after medication
(AUClast) | 0~144 hour after medication

SECONDARY OUTCOMES:
(AUCinf) | 0~144 hour after medication
(tmax) | 0~144 hour after medication
(t1/2) | 0~144 hour after medication

CONTACTS AND LOCATIONS:
Overall Officials: seunghoon han, M.D., Ph.D., Principal Investigator — The Catholic university St. Mary hospital
Locations (1):
- The Catholic university St. Mary hospital, Seoul, South Korea